CLINICAL TRIAL: NCT07012967
Title: Effects of Thoracic Kinesio Taping on Pulmonary Function, Respiratory Muscle Strength, and Sleep Quality in Obese and Overweight Individuals
Brief Title: Kinesio Taping in Obesity: Breathing and Sleep Implications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Kabasakal (Other)
Responsible Party: Sponsor-Investigator, Elif Kabasakal, LECTURER, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISU-2025-004
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: obesity; Kinesio taping; respiratory function; sleep
MeSH Terms: conditions — Obesity; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping (Experimental): Thoracic kinesiology taping will be applied using 5 cm-wide, latex-free cotton tape following Kase's
  Interventions: Other: Kinesiology Taping
- control group (Other): Participants in the control group will receive diaphragmatic breathing exercises. Exercises will be taught and supervised by a physiotherapist. Sessions will be conducted twice weekly for four weeks, and participants will be instructed to continue home practice between sessions.
  Interventions: Other: Diaphragmatic Breathing Exercises

INTERVENTIONS:
Other: Kinesiology Taping — For thoracic kinesiology taping (KT), a 5 cm wide, 100% cotton, latex-free elastic tape will be used. Application sites will follow the technique and principles described by Kase. Participants will sit upright in an armless chair with knees at 90° flexion, feet flat on the floor, and arms relaxed.
  The tape will be applied to the front and back of the body to facilitate respiratory muscles, primarily the diaphragm. On the anterior side, an "I"-shaped strip will be applied with 50-75% tension at the xiphoid process along the linea alba, and the tails will be laid over the subcostal area without tension. Posteriorly, another "I"-shaped strip will be applied from the projection of the 12th thoracic vertebra with 50-75% tension, and the ends placed toward the ribs without tension. Additionally, two more strips will be applied to the upper trapezius region between the neck and acromion bilaterally.
  Arms: Kinesiology Taping
Other: Diaphragmatic Breathing Exercises — Participants in the control group will receive diaphragmatic breathing exercises. Exercises will be taught and supervised by a physiotherapist. Sessions will be conducted twice weekly for four weeks, and participants will be instructed to continue home practice between sessions.
  Arms: control group

SUMMARY:
Obesity, defined as excessive fat accumulation, is a chronic, complex, and global health issue. It is increasingly prevalent worldwide and is considered a disease that requires treatment. According to recent data, 43% of adults aged 18 and over were classified as overweight, and 16% as obese. In Turkey, a national health survey reported that among individuals aged 15 and above, 20.2% were obese, and 35.6% were in a pre-obese state based on their body mass index (BMI).

The effects of excess weight on health are significant, as weight gain shortens life expectancy and reduces quality of life. Obesity has detrimental effects on many systems, including the respiratory system. It reduces the compliance of the lungs and chest wall, alters respiratory patterns and ventilation-perfusion relationships, impairs gas exchange, and decreases lung volumes. In some individuals, respiratory control is altered due to the effects of adipokines, which can lead to hypoventilation and increased levels of carbon dioxide in the blood (hypercapnia).

Obesity affects the respiratory system both symptomatically (e.g., shortness of breath) and functionally. Respiratory function disorders in individuals with obesity may include decreased functional residual capacity (FRC), expiratory reserve volume (ERV), and, in some cases, reduced total lung capacity (TLC). Additionally, obesity is a health issue that affects sleep quality. There are three proposed bidirectional relationships: obesity causes poor sleep, poor sleep contributes to obesity, and both may coexist. Individuals with obesity often report poor sleep quality and sleep disorders such as sleep apnea.

The primary function of the respiratory system is gas exchange, which is closely related to the mechanical properties of the respiratory pump. The functionality of this pump depends on the interaction of the lungs, abdominal wall, ribs, intercostal muscles, and the diaphragm. In diseases that impair the structure of the diaphragm, improving its function can alleviate symptoms and significantly enhance pulmonary function test results.

Kinesiology taping (KT), an elastic therapeutic taping method, is commonly used for musculoskeletal disorders but has a wide range of clinical applications. Kinesiology tapes are reported to support weak muscles, increase circulation, reduce pain by stimulating the neurological system, provide proprioceptive feedback, and correct joint misalignments. The mechanism by which KT influences muscle strength depends on the application technique, which can either enhance or inhibit muscle activation. The underlying mechanism is explained by the stimulation of sensory-motor and proprioceptive systems, aiming to improve muscle function through enhanced neuromuscular feedback. Kinesiology taping has also shown potential benefits in respiratory conditions by improving diaphragm function, reducing respiratory muscle fatigue, and enhancing overall respiratory mechanics.

Understanding the effects of thoracic kinesiology taping on respiratory function, vital signs, sleep, quality of life, and cognitive functions in individuals with obesity is of great importance for physiotherapists and researchers. The findings from this study may provide valuable insights for developing comprehensive rehabilitation programs and improving the health status of individuals with obesity. Therefore, the aim of this study is to investigate the effects of thoracic kinesiology taping on respiratory functions, respiratory muscle strength, vital signs, sleep, quality of life, and cognitive status in individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 70 years of age
* Being overweight or classified as class 1 or class 2 obese based on BMI
* Having the ability to follow instructions and participate in study procedures
* Being able to speak and understand Turkish

Exclusion Criteria:

* Having an acute or chronic pulmonary or respiratory disease
* Having an uncontrolled chronic illness
* Having an allergic reaction to kinesiology tape
* Refusing to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | At baseline (before the intervention) and at the end of the 4th week of intervention
  Forced Vital Capacity (FVC) will be measured using a portable spirometer (Cosmed Pony FX, Italy) following ATS/ERS guidelines. Results will be recorded in liters and as a percentage of the predicted value.
Forced Expiratory Volume in 1 Second (FEV1) | At baseline (before the intervention) and at the end of the 4th week of intervention
  FEV1 will be assessed using a spirometer (Cosmed Pony FX) under ATS/ERS standards. The measurement will be recorded in liters and as a percentage of the predicted normal value.
FEV1/FVC Ratio | At baseline (before the intervention) and at the end of the 4th week of intervention
  The ratio of FEV1 to FVC (FEV1/FVC) will be calculated to assess airway obstruction. The values will be expressed as a percentage. All procedures will be carried out with standardized spirometry protocols (ATS/ERS) using single-use mouthpieces and filters.
Peak Expiratory Flow (PEF) | At baseline (before the intervention) and at the end of the 4th week of intervention
  PEF will be measured as part of the pulmonary function test using a spirometer. Values will be expressed in liters per second (L/s) and as a percentage of the predicted value. Infection control procedures will include the use of disposable mouthpieces and filters as per device guidelines.
Maximal Inspiratory Pressure (MIP) | Baseline and Week 4 (Post-Intervention)
  Maximal Inspiratory Pressure (MIP) will be measured using a portable electronic mouth pressure device (Micro Medical Micro RPM, UK). The measurement will be performed during maximal inspiratory effort against an occluded airway after full expiration and held for 1-3 seconds. Three trials will be conducted, and the highest value will be recorded. Results will be expressed in cmH₂O and as a percentage of age- and sex-predicted reference values. Infection control procedures will include disposable, single-use mouthpieces and filters.
Maximal Expiratory Pressure (MEP) | Baseline and Week 4 (Post-Intervention)
  Maximal Expiratory Pressure (MEP) will be assessed using a portable electronic mouth pressure device (Micro Medical Micro RPM, UK). The participant will first perform maximal inspiration, then exhale maximally against an occluded airway for 1-3 seconds. The best of three measurements will be used. Data will be reported in cmH₂O and as a percentage of predicted values based on age and sex. Standard infection control measures with single-use mouthpieces and filters will be followed.
Pittsburgh Sleep Quality Index (PSQI) Total Score | Baseline and Week 4 (Post-Intervention)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-report questionnaire consisting of 19 items grouped into 7 components. Each item is scored from 0 to 3, and the sum of the 7 component scores yields a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality. A total score of ≤5 indicates good sleep quality, while >5 indicates poor sleep quality. The validated Turkish version will be used in this study.

SECONDARY OUTCOMES:
Heart Rate (HR) | Baseline, Week 4 (Post-Intervention), and Daily During Weeks 1-4
  Heart rate (HR) will be measured in beats per minute (bpm) using a validated digital pulse oximeter or heart rate monitor. Measurements will be taken at baseline and at the end of the 4th week, as well as daily during the intervention period (upon waking, during the day, and before sleep).
Oxygen Saturation (SpO₂) | Baseline, Week 4 (Post-Intervention), and Daily During Weeks 1-4
  Peripheral oxygen saturation (SpO₂) will be assessed using a digital pulse oximeter. Measurements will be recorded as a percentage and monitored daily during the intervention period, including morning, daytime, and pre-sleep values, along with baseline and end-of-intervention readings.
Blood Pressure (Systolic and Diastolic) | Baseline, Week 4 (Post-Intervention), and Daily During Weeks 1-4
  Systolic and diastolic blood pressure (BP) will be measured in mmHg using an automated upper-arm digital sphygmomanometer. Readings will be obtained at baseline and at the end of Week 4, as well as daily throughout the intervention (morning, daytime, and before bedtime).
Obesity-Specific Quality of Life Questionnaire (OQOLQ) Total Score | Baseline and Week 4 (Post-Intervention)
  Obesity-specific quality of life will be assessed using the OQOLQ, a validated 17-item scale developed by Patrick et al. Each item is scored on a six-point Likert scale. The scale is unidimensional, and higher total scores indicate poorer quality of life. The validated Turkish version will be used in this study.
Auditory-Visual Number Sequence Test (GİSDT) Total Score | Baseline and Week 4 (Post-Intervention)
  Cognitive function, particularly short-term memory, attention, and concentration, will be assessed using the Auditory-Visual Number Sequence Test (GİSDT). The test includes four subtests: Auditory-Verbal, Visual-Verbal, Auditory-Written, and Visual-Written. Participants are presented with number sequences that increase in length, either by hearing or seeing them, and are required to repeat them in the same order, either verbally or in writing. The score reflects the longest sequence correctly recalled without error in one of two attempts. The Turkish standardized version will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Istınye University, Istanbul,, Istanbul, Turkey (Türkiye)